CLINICAL TRIAL: NCT05305001
Title: Prevalence Estimation of BRCA1, BRCA2 and Other Germline Mutations Associated With Hereditary Pancreatic Cancer Using a Comprehensive Gene Panel in an Unselected Cohort of Patients With Pancreatic Adenocarcinoma in Mexico
Brief Title: Germline Mutations Associated With Hereditary Pancreatic Cancer in Unselected Patients With Pancreatic Cancer in Mexico
Status: Completed | Type: Observational
Sponsor: Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran (Other)
Responsible Party: Sponsor
Other Study IDs: HEM-3331-20-20-1
Record Dates: First submitted 2021-06-02; First posted 2022-03-31 (Actual); Last update posted 2022-10-18 (Actual); Status verified 2022-10

CONDITIONS: Pancreatic Cancer; Pancreatic Adenocarcinoma
Keywords: BRCA 1/2 germline mutations
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 5 mL of whole blood mixed with EDTA will be collected from each participant.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Genetic: Invitae Multi-Cancer Panel ® — Participants will have genetic testing.

SUMMARY:
Pancreatic cancer is a highly lethal disease. The cause of pancreatic cancer is multifactorial. However, around 10% of cases are associated with hereditary predisposition. Germline mutations in BRCA1 and BRCA2, CDKN2A, STK11, DNA mismatch repair (MMR) genes (MLH1, MSH2, MSH6, or PMS2), PALB2, FANCC, FANCG, and ATM have been associated with an increased risk for pancreatic cancer. The prevalence of these germline mutations varies across populations. For instance, the prevalence of BRCA1/2 germline mutations in high-risk populations can be up to 20%. On the other hand, in unselected patient population, the prevalence of BRCA1/2 germline mutations is 5-7%. In Mexican population, data on the prevalence of BRCA1/2 germline mutations in patients with pancreatic cancer are lacking. Identification of BRCA germline mutations in patients with pancreatic cancer has implications for treatment. Also, it allows genetic testing and counselling for family members. This study will determine the prevalence of germline mutations associated with hereditary pancreatic cancer using a comprehensive gene panel in an unselected cohort of patients with pancreatic adenocarcinoma in Mexico.

DETAILED DESCRIPTION:
This is an observational study to estimate the prevalence of germline mutations in patients with pancreatic cancer. Eighty four genes will be analyzed, all of which have been associated with hereditary cancer. The genes are included on Invitae Multi-Cancer Panel ®, performing full-gene sequencing and deletion/duplication analysis using next-generation sequencing technology. The 84 genes include: AIP, ALK, APC, ATM, AXIN2, BAP1, BARD1, BLM, BMPR1A, BRCA1, BRCA2, BRIP1, CASR, CDC73, CDH1, CDK4, CDKN1B, CDKN1C, CDKN2A, CEBPA, CHEK2, CTNNA1, DICER1, DIS3L2, EGFR, EPCAM, FH, FLCN, GATA2, GPC3, GREM1, HOXB13, HRAS, KIT, MAX, MEN1, MET, MITF, MLH1, MSH2, MSH3, MSH6, MUTYH, NBN, NF1, NF2, NTHL1, PALB2, PDGFRA, PHOX2B, PMS2, POLD1, POLE, POT1, PRKAR1A, PTCH1, PTEN, RAD50, RAD51C, RAD51D, RB1, RECQL4, RET, RUNX1, SDHA, SDHAF2, SDHB, SDHC, SDHD, SMAD4, SMARCA4, SMARCB1, SMARCE1, STK11, SUFU, TERC, TERT, TMEM127, TP53, TSC1, TSC2, VHL, WRN, WT1.

ELIGIBILITY:
Inclusion Criteria:

* Female and male participants ≥ 18 years of age.
* Diagnosed within the previous 6 months with histologically confirmed pancreatic adenocarcinoma stage I to IV.
* Participant provides written informed consent for the study.
* Participant must agree to sample collection and genetic testing using the Invitae Multi-Cancer Panel ®.

Exclusion Criteria:

* Diagnosed with pancreatic adenocarcinoma more than 6 months before presenting to the clinical site.
* Diagnosed with intraductal papillary mucinous neoplasms, mucinous cystic neoplasms, pancreatic neuroendocrine tumors.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be patients who are diagnosed within 6 months of enrollment with pancreatic adenocarcinoma.
Sampling Method: Probability Sample
Enrollment: 107 (Actual)
Dates: Start 2020-09-09 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
BRCA 1/2 germline mutation prevalence | 15 months
  To estimate the prevalence of BRCA1 and BRCA2 germline mutations in patients who present to the clinical site within 6 months of a histologically confirmed diagnosis of pancreatic adenocarcinoma.

SECONDARY OUTCOMES:
Other germline mutation prevalence | 15 months
  To estimate the prevalence of other germline mutations associated with hereditary pancreatic cancer in patients who present to the clinical site within 6 months of a histologically confirmed diagnosis of pancreatic adenocarcinoma.
Clinical and pathological characteristics | 15 months
  To describe the clinical and pathological characteristics of patients with pancreatic adenocarcinoma and BRCA1, BRCA2 and other germline mutations.

OTHER OUTCOMES:
The proportion of blood relatives of germline mutation carriers who accept genetic counseling and genetic testing | 15 months
  Number of first degree relatives with a positive genetic test result. Number of first degree relatives with genetic counseling and genetic testing.
The proportion of germline mutation carriers who accept pancreatic cancer surveillance. | up to 15 months
  Number of germline mutation carriers included in a surveillance protocol assessed by abdominal imaging.

CONTACTS AND LOCATIONS:
Overall Officials: Fidel D Huitzil Meléndez, MD, Principal Investigator — Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran
Locations (1):
- Instituto Nacional de Ciencias Médicas y Nutrición Salvador Zubirán, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bray F, Ferlay J, Soerjomataram I, Siegel RL, Torre LA, Jemal A. Global cancer statistics 2018: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2018 Nov;68(6):394-424. doi: 10.3322/caac.21492. Epub 2018 Sep 12. PMID 30207593
- [Background] Rawla P, Sunkara T, Gaduputi V. Epidemiology of Pancreatic Cancer: Global Trends, Etiology and Risk Factors. World J Oncol. 2019 Feb;10(1):10-27. doi: 10.14740/wjon1166. Epub 2019 Feb 26. PMID 30834048
- [Background] Hruban RH, Canto MI, Goggins M, Schulick R, Klein AP. Update on familial pancreatic cancer. Adv Surg. 2010;44:293-311. doi: 10.1016/j.yasu.2010.05.011. No abstract available. PMID 20919528
- [Background] Venkitaraman AR. Cancer suppression by the chromosome custodians, BRCA1 and BRCA2. Science. 2014 Mar 28;343(6178):1470-5. doi: 10.1126/science.1252230. PMID 24675954
- [Background] Gorodetska I, Kozeretska I, Dubrovska A. BRCA Genes: The Role in Genome Stability, Cancer Stemness and Therapy Resistance. J Cancer. 2019 May 14;10(9):2109-2127. doi: 10.7150/jca.30410. eCollection 2019. PMID 31205572
- [Background] Murphy KM, Brune KA, Griffin C, Sollenberger JE, Petersen GM, Bansal R, Hruban RH, Kern SE. Evaluation of candidate genes MAP2K4, MADH4, ACVR1B, and BRCA2 in familial pancreatic cancer: deleterious BRCA2 mutations in 17%. Cancer Res. 2002 Jul 1;62(13):3789-93. PMID 12097290
- [Background] Stadler ZK, Salo-Mullen E, Patil SM, Pietanza MC, Vijai J, Saloustros E, Hansen NA, Kauff ND, Kurtz RC, Kelsen DP, Offit K, Robson ME. Prevalence of BRCA1 and BRCA2 mutations in Ashkenazi Jewish families with breast and pancreatic cancer. Cancer. 2012 Jan 15;118(2):493-9. doi: 10.1002/cncr.26191. Epub 2011 May 19. PMID 21598239
- [Background] Risch HA, McLaughlin JR, Cole DE, Rosen B, Bradley L, Fan I, Tang J, Li S, Zhang S, Shaw PA, Narod SA. Population BRCA1 and BRCA2 mutation frequencies and cancer penetrances: a kin-cohort study in Ontario, Canada. J Natl Cancer Inst. 2006 Dec 6;98(23):1694-706. doi: 10.1093/jnci/djj465. PMID 17148771
- [Background] Fernandez-Lopez JC, Romero-Cordoba S, Rebollar-Vega R, Alfaro-Ruiz LA, Jimenez-Morales S, Beltran-Anaya F, Arellano-Llamas R, Cedro-Tanda A, Rios-Romero M, Ramirez-Florencio M, Bautista-Pina V, Dominguez-Reyes C, Villegas-Carlos F, Tenorio-Torres A, Hidalgo-Miranda A. Population and breast cancer patients' analysis reveals the diversity of genomic variation of the BRCA genes in the Mexican population. Hum Genomics. 2019 Jan 10;13(1):3. doi: 10.1186/s40246-018-0188-9. PMID 30630528
- [Background] Villarreal-Garza C, Alvarez-Gomez RM, Perez-Plasencia C, Herrera LA, Herzog J, Castillo D, Mohar A, Castro C, Gallardo LN, Gallardo D, Santibanez M, Blazer KR, Weitzel JN. Significant clinical impact of recurrent BRCA1 and BRCA2 mutations in Mexico. Cancer. 2015 Feb 1;121(3):372-8. doi: 10.1002/cncr.29058. Epub 2014 Sep 18. PMID 25236687
- [Background] Villarreal-Garza C, Weitzel JN, Llacuachaqui M, Sifuentes E, Magallanes-Hoyos MC, Gallardo L, Alvarez-Gomez RM, Herzog J, Castillo D, Royer R, Akbari M, Lara-Medina F, Herrera LA, Mohar A, Narod SA. The prevalence of BRCA1 and BRCA2 mutations among young Mexican women with triple-negative breast cancer. Breast Cancer Res Treat. 2015 Apr;150(2):389-94. doi: 10.1007/s10549-015-3312-8. Epub 2015 Feb 26. PMID 25716084
- [Background] Golan T, Hammel P, Reni M, Van Cutsem E, Macarulla T, Hall MJ, Park JO, Hochhauser D, Arnold D, Oh DY, Reinacher-Schick A, Tortora G, Algul H, O'Reilly EM, McGuinness D, Cui KY, Schlienger K, Locker GY, Kindler HL. Maintenance Olaparib for Germline BRCA-Mutated Metastatic Pancreatic Cancer. N Engl J Med. 2019 Jul 25;381(4):317-327. doi: 10.1056/NEJMoa1903387. Epub 2019 Jun 2. PMID 31157963
- See also: globocan — http://gco.iarc.fr

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2020-07-20): https://cdn.clinicaltrials.gov/large-docs/01/NCT05305001/Prot_SAP_ICF_000.pdf